CLINICAL TRIAL: NCT03767452
Title: A Phase 4, Single-Center, Multiple-Dose, Open-Label Trial to Evaluate the Efficacy of Additional Xiaflex® Treatment in Patients With Peyronie's Disease Recurrence, Worsening, or Incomplete Response After Prior Xiaflex® Treatment
Brief Title: Additional Xiaflex® Treatment in Patients With Peyronie's Disease Recurrence, Worsening, or Incomplete Response
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manhattan Medical Research Practice, PLLC (Industry)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMR032018
Record Dates: First submitted 2018-11-30; First posted 2018-12-06 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Peyronie's Disease
Keywords: Recurrence; Incomplete Response; Worsening; Curvature
MeSH Terms: conditions — Penile Induration; Recurrence | interventions — Microbial Collagenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single-Arm (Experimental): Xiaflex® 0.58 mg, 2 injections separated by 1 to 3 days, repeated after 6 weeks for up to 4 treatment cycles.
  Interventions: Drug: Xiaflex® 0.58 mg

INTERVENTIONS:
Drug: Xiaflex® 0.58 mg — 0.25 mL injections.

SUMMARY:
Subjects who have had an incomplete response to previous Xiaflex® will receive up to 4 additional cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent to participate in the study.
2. Male aged ≥18 years old at screening.
3. Previously received Xiaflex® treatment and had a partial or complete response.

   * Partial response is defined as receiving ≤ 4 cycles of Xiaflex® and achieving a penile curvature of ≥ 15 degrees and < 90 degrees.
   * Complete response is defined as receiving ≤ 4 cycles of Xiaflex® and achieving a penile curvature of < 15 degrees.
4. Has a diagnosis of Peyronie's disease with a penile curvature of ≥ 30 and ≤ 90 degrees at the screening visit.
5. Has a penile curvature of at ≥ 30 degrees in the dorsal, lateral, or dorsal/lateral plane at the screening visit. It must be possible to delineate the single plane of maximal curvature for evaluation during the study.
6. Able and willing to comply with restrictions where intercourse or any other sexual activity is prohibited during each treatment cycle and for at least 2 weeks after each injection cycle.
7. Able and willing to perform home modeling sessions between injection cycles.
8. Is in good health based on medical history evaluation and in the judgment of the principal investigator.

Exclusion Criteria:

1. Has a penile curvature of < 30 degrees or > 90 degrees at the screening visit.
2. Previous allergic reaction to XIAFLEX®.
3. Has any of the following conditions:

   * Chordee in the presence or absence of hypospadias
   * Thrombosis of the dorsal penile artery and or vein
   * Infiltration by a benign or malignant mass resulting in penile curvature
   * Infiltration by an infectious agent, such as lymphogranuloma venereum
   * Ventral curvature from any cause
   * Presence of an active sexually transmitted disease
   * Known active hepatitis B or C
   * Known human immune deficiency virus (HIV)
4. Has previously undergone surgery for Peyronie's disease.
5. Has an erection which, in the opinion of the investigator, is insufficient to accurately measure the subject's penile deformity after administration of the prostaglandin E1 (PGE1), Trimix®, or similar erection inducing agent.
6. Has a calcified plaque that, in the opinion of the investigator, would prevent proper administration of the study medication.
7. Has an isolated hourglass deformity of the penis.
8. Has a plaque causing a curvature of the penis located proximal to the base of the penis where injection of local anesthetic would interfere with the injection of Xiaflex®.
9. Has received intralesional or injection therapy for Peyronie's disease including interferon, verapamil, or Xiaflex® < 6 months prior to screening.
10. Has used antiplatelet or anti-coagulants (e.g. coumadin, Plavix®, Eliquis®, Effient®) within 7 days prior to each Xiaflex® injection. Daily aspirin of 81 mg is acceptable.
11. Has had extracorporeal shock wave therapy (ESWT) for the correction of Peyronie's disease within the 6 months prior to screening or plans to have ESWT at any time during the study.
12. Has uncontrolled hypertension as determined by the investigator.
13. Has a recent history of stroke, bleeding, or other significant medical condition which, in the investigator's opinion, would make the subject unsuitable for enrollment in the study.
14. Has a planned surgical procedure during anticipated study participation.
15. Is unwilling or unable to cooperate with the requirements of the study including completion of all scheduled study visits.
16. Has received investigational drug or treatment within 30 days of the first dose Xiaflex®.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Change in the degree of penile curvature | From Screening up to 24 weeks
  Measurable change in the curvature of penis

CONTACTS AND LOCATIONS:
Overall Officials: Jed Kaminetsky, MD, Principal Investigator — Principal Investigator
Locations (1):
- Manhattan Medical Research Practice, PLLC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided